CLINICAL TRIAL: NCT03810703
Title: Hypomania, Amphetamine, and Preferences for Sweets
Brief Title: Differential Responses to Drugs and Sweet Tastes
Acronym: HAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB16-1293
Record Dates: First submitted 2017-08-01; First posted 2019-01-22 (Actual); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-05

CONDITIONS: Bipolar II Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Dextroamphetamine

STUDY DESIGN:
Intervention Model Description: Study will track participants in two assigned groups (participants that exhibit either High or Low Bipolar II/Hypomanic phenotypes)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- placebo arm (Placebo Comparator): Participant will receive placebo oral capsule during this four hour session.
  Interventions: Drug: Placebo oral capsule
- amphetamine 10 mg arm (Experimental): Participant will receive d-amphetamine 10 mg oral capsule during this four hour session.
  Interventions: Drug: d-amphetamine 10 mg oral capsule
- amphetamine 20 mg arm (Experimental): Participant will receive d-amphetamine 20 mg oral capsule during this four hour session.
  Interventions: Drug: d-amphetamine 20 mg oral capsule

INTERVENTIONS:
Drug: Placebo oral capsule — Placebo oral capsule
  Arms: placebo arm
Drug: d-amphetamine 10 mg oral capsule — d-amphetamine 10 mg oral capsule
  Arms: amphetamine 10 mg arm
Drug: d-amphetamine 20 mg oral capsule — d-amphetamine 20 mg oral capsule
  Arms: amphetamine 20 mg arm

SUMMARY:
Young adults who exhibit "bipolar phenotype" (BPP), defined as occasional episodes of mood elevation and heightened activity, are at risk for several psychiatric disorders, including problem use of drugs and alcohol. Mood elevation has been linked to higher alcohol consumption and alcohol use disorders. Individuals with BPP show elevated lifetime prevalence of alcohol use disorders (between 39%-61%), figures that exceed those reported in both major depression and schizophrenia. Recently, the investigators demonstrated in a controlled laboratory study that individuals with BPP (but not meeting criteria for full Bipolar I Disorder), report dampened responses to a single dose of alcohol, compared to placebo. In the current study, the investigators seek to extend these findings to determine if young adults reporting BPP, based on a questionnaire, will exhibit reduced responses to other rewarding stimuli, such as d-amphetamine and sweet tastes. The investigators hypothesize that the BPP individuals will exhibit dampened subjective responses to stimulant and sweet taste rewards compared to healthy controls.

DETAILED DESCRIPTION:
This study will extend the understanding of risk factors for drug or alcohol misuse, or other reward-related behaviors. The investigators previously showed that individuals who report occasional feelings of high energy and excitability experience less effect from a single dose of alcohol, compared to people who have not experienced these effects. Now the investigators wish to determine if this dampened response also occurs with other rewards, namely feelings of wellbeing after a dose of amphetamine, or liking of a sweet solution. Individuals who exhibit the BPP (i.e., periods of excitability) also are more likely to develop alcohol problems, substance misuse, and weight gain and obesity. Therefore, the investigators will test the working hypothesis that young adults who report having these experiences, based on a questionnaire measure (i.e., BPP individuals) will show dampened subjective responses to both single oral doses of amphetamine or sweet palatable tastes. The investigators will also obtain objective measures (e.g. Respiratory Sinus Arrhythmia and heart rate) to amphetamine and sweet taste, to establish whether the dampened subjective response extends to physiological indices as well. This study will extend the previous literature regarding the blunted effects of alcohol in BPP individuals and will suggest possible mechanisms that promote broader addictive behaviors in individuals with mood disturbance. Importantly, the investigators are proposing to test individuals at a relatively young age, 18-19 years. This is important to identify a risk factor, that is thought to pre-date use of drugs. In older participants, it would be difficult to separate the role of the pre-existing trait from the effect of habitual drug or alcohol use that escalates markedly after age 20.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-19 years old
* BMI of 19-26
* Physical/EKG/Medical History/Medications Approved by Physician for d-amphetamine
* at least High School education
* Fluent in English

Exclusion Criteria:

* No Current Mood, Anxiety, Eating or Psychotic Disorder
* No current psychotropic medication
* No Recent Drug Dependence
* < 4 alcoholic drinks/day for males; < 3 alcoholic drinks/day for females (monthly average)
* No weekly (or more frequent) illicit drug use
* No women who are pregnant, nursing, or planning pregnancy within 3 months (birth control is okay)

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Chicago Medical Center - Human Behavioral Pharmacology Lab, Chicago, Illinois
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calabrese JR, Hirschfeld RM, Reed M, Davies MA, Frye MA, Keck PE, Lewis L, McElroy SL, McNulty JP, Wagner KD. Impact of bipolar disorder on a U.S. community sample. J Clin Psychiatry. 2003 Apr;64(4):425-32. doi: 10.4088/jcp.v64n0412. PMID 12716245
- [Background] Chandler RA, Wang PW, Ketter TA, Goodwin GM. A new US-UK diagnostic project: mood elevation and depression in first-year undergraduates at Oxford and Stanford universities. Acta Psychiatr Scand. 2008 Jul;118(1):81-5. doi: 10.1111/j.1600-0447.2008.01193.x. PMID 18595178
- [Background] de Lauzon B, Romon M, Deschamps V, Lafay L, Borys JM, Karlsson J, Ducimetiere P, Charles MA; Fleurbaix Laventie Ville Sante Study Group. The Three-Factor Eating Questionnaire-R18 is able to distinguish among different eating patterns in a general population. J Nutr. 2004 Sep;134(9):2372-80. doi: 10.1093/jn/134.9.2372. PMID 15333731
- [Background] Francis LJ, Robbins M, Louden SH, Haley JM. A revised psychoticism scale for the revised Eysenck personality questionnaire: a study among clergy. Psychol Rep. 2001 Jun;88(3 Pt 2):1131-4. doi: 10.2466/pr0.2001.88.3c.1131. PMID 11597066
- [Background] Williams JB, Gibbon M, First MB, Spitzer RL, Davies M, Borus J, Howes MJ, Kane J, Pope HG Jr, Rounsaville B, et al. The Structured Clinical Interview for DSM-III-R (SCID). II. Multisite test-retest reliability. Arch Gen Psychiatry. 1992 Aug;49(8):630-6. doi: 10.1001/archpsyc.1992.01820080038006. PMID 1637253
- [Background] Grossman P, Taylor EW. Toward understanding respiratory sinus arrhythmia: relations to cardiac vagal tone, evolution and biobehavioral functions. Biol Psychol. 2007 Feb;74(2):263-85. doi: 10.1016/j.biopsycho.2005.11.014. Epub 2006 Nov 1. PMID 17081672
- [Background] Grossman P, van Beek J, Wientjes C. A comparison of three quantification methods for estimation of respiratory sinus arrhythmia. Psychophysiology. 1990 Nov;27(6):702-14. doi: 10.1111/j.1469-8986.1990.tb03198.x. PMID 2100356
- [Background] Haertzen CA. Development of scales based on patterns of drug effects, using the addiction Research Center Inventory (ARCI). Psychol Rep. 1966 Feb;18(1):163-94. doi: 10.2466/pr0.1966.18.1.163. No abstract available. PMID 5908477
- [Background] Hoeppner BB, Stout RL, Jackson KM, Barnett NP. How good is fine-grained Timeline Follow-back data? Comparing 30-day TLFB and repeated 7-day TLFB alcohol consumption reports on the person and daily level. Addict Behav. 2010 Dec;35(12):1138-43. doi: 10.1016/j.addbeh.2010.08.013. Epub 2010 Aug 13. PMID 20822852
- [Background] Hirschfeld RM, Holzer C, Calabrese JR, Weissman M, Reed M, Davies M, Frye MA, Keck P, McElroy S, Lewis L, Tierce J, Wagner KD, Hazard E. Validity of the mood disorder questionnaire: a general population study. Am J Psychiatry. 2003 Jan;160(1):178-80. doi: 10.1176/appi.ajp.160.1.178. PMID 12505821
- [Background] Waleeprakhon P, Ittasakul P, Lotrakul M, Wisajun P, Jullagate S, Ketter TA. Development and validation of a screening instrument for bipolar spectrum disorder: The Mood Disorder Questionnaire Thai version. Neuropsychiatr Dis Treat. 2014 Aug 18;10:1497-502. doi: 10.2147/NDT.S67842. eCollection 2014. PMID 25170269
- [Background] Jacob T, Seilhamer RA, Bargeil K, Howell DN. Reliability of Lifetime Drinking History among alcohol dependent men. Psychol Addict Behav. 2006 Sep;20(3):333-7. doi: 10.1037/0893-164X.20.3.333. PMID 16938072
- [Background] Johanson CE, Uhlenhuth EH. Drug preference and mood in humans: d-amphetamine. Psychopharmacology (Berl). 1980;71(3):275-9. doi: 10.1007/BF00433062. PMID 6779335
- [Background] Kessler RC, Crum RM, Warner LA, Nelson CB, Schulenberg J, Anthony JC. Lifetime co-occurrence of DSM-III-R alcohol abuse and dependence with other psychiatric disorders in the National Comorbidity Survey. Arch Gen Psychiatry. 1997 Apr;54(4):313-21. doi: 10.1001/archpsyc.1997.01830160031005. PMID 9107147
- [Background] Regier DA, Farmer ME, Rae DS, Locke BZ, Keith SJ, Judd LL, Goodwin FK. Comorbidity of mental disorders with alcohol and other drug abuse. Results from the Epidemiologic Catchment Area (ECA) Study. JAMA. 1990 Nov 21;264(19):2511-8. PMID 2232018
- [Background] Rock PL, Goodwin GM, Harmer CJ. The common adolescent bipolar phenotype shows positive biases in emotional processing. Bipolar Disord. 2010 Sep;12(6):606-15. doi: 10.1111/j.1399-5618.2010.00859.x. PMID 20868459
- [Background] Trost S, Diekhof EK, Mohr H, Vieker H, Kramer B, Wolf C, Keil M, Dechent P, Binder EB, Gruber O. Investigating the Impact of a Genome-Wide Supported Bipolar Risk Variant of MAD1L1 on the Human Reward System. Neuropsychopharmacology. 2016 Oct;41(11):2679-87. doi: 10.1038/npp.2016.70. Epub 2016 May 13. PMID 27184339
- [Background] Weafer J, Burkhardt A, de Wit H. Sweet taste liking is associated with impulsive behaviors in humans. Front Behav Neurosci. 2014 Jun 17;8:228. doi: 10.3389/fnbeh.2014.00228. eCollection 2014. PMID 24987343
- [Background] Gontkovsky ST. Sensitivity of the Wechsler Abbreviated Scale of Intelligence-Second Edition (WASI-II) to the neurocognitive deficits associated with the semantic dementia variant of frontotemporal lobar degeneration: A case study. Appl Neuropsychol Adult. 2017 May-Jun;24(3):288-293. doi: 10.1080/23279095.2016.1154857. Epub 2016 Apr 21. PMID 27101084
- [Background] White TL, Justice AJ, de Wit H. Differential subjective effects of D-amphetamine by gender, hormone levels and menstrual cycle phase. Pharmacol Biochem Behav. 2002 Nov;73(4):729-41. doi: 10.1016/s0091-3057(02)00818-3. PMID 12213517
- [Background] Yip SW, Doherty J, Wakeley J, Saunders K, Tzagarakis C, de Wit H, Goodwin GM, Rogers RD. Reduced subjective response to acute ethanol administration among young men with a broad bipolar phenotype. Neuropsychopharmacology. 2012 Jul;37(8):1808-15. doi: 10.1038/npp.2012.45. Epub 2012 Apr 11. PMID 22491350

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Arm | Amphetamine 10 mg Arm | Amphetamine 20 mg Arm
Started | 31 | 31 | 31
Completed | 31 | 31 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Amphetamine 10 mg Arm | Amphetamine 20 mg Arm | Total
Number analyzed (Participants) | 31 | 31 | 31 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 31 | 31 | 93
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 13 | 39
  Male | 18 | 18 | 18 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 4 | 12
  White | 24 | 24 | 24 | 72
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 31 | 93
Education - High School Education [Count of Participants; unit: Participants] | 31 | 31 | 31 | 93

OUTCOME MEASURES:

1. Primary Outcome: Change in Subjective Effects as Assessed by Score on "Feel Drug", "Feel High", "Like Drug", and "Want More" Sub-scales of Drug Effects Questionnaire (DEQ).
Description: Participants will complete The Drug Effects Questionnaire during the initial baseline session to determine their subjective stimulant profile. The Dug Effects Questionnaire (DEQ) is a visual analog scale questionnaire that assesses the extent to which subjects experience four subjective states: "Feel Drug", "Feel High", "Like Drug", and "Want More". All sub-scales are scored on a visual analogue scale (Scroll bar on computer screen) ranging from 0-100. 100 represents the highest score for that subjective state, and the higher the score, the worse the outcome.
Time Frame: End of study (Baseline - time 0 and approximately 4 weeks later)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Arm | Amphetamine 10 mg Arm | Amphetamine 20 mg Arm
Number analyzed (Participants) | 31 | 31 | 31
score on a scale
  Feel | 18.88 (8.84) | 35.25 (4.46) | 45.75 (8.23)
  Like | 37.44 (7.64) | 50.69 (7.82) | 52.81 (8.96)
  Dislike | 19.00 (5.96) | 27.19 (6.47) | 16.25 (5.15)
  High | 17.50 (5.50) | 24.88 (5.48) | 32.69 (8.68)
  More | 29.19 (7.56) | 45.38 (7.66) | 52.44 (8.40)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 5 weeks
Arm/Group | Placebo Arm | Amphetamine 10 mg Arm | Amphetamine 20 mg Arm
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT03810703/Prot_SAP_000.pdf